CLINICAL TRIAL: NCT04967807
Title: Myocardial Injury and Outcomes Following COVID-19 Vaccination (MYOVAX Study)
Acronym: MYOVAX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-5621
Record Dates: First submitted 2021-06-29; First posted 2021-07-20 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Myocardial Injury; Myocarditis; COVID-19 Vaccination; SARS-CoV-2; Cardiac MRI
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Intervention Model Description: The study population will include 2 cohorts of patients post COVID-19 vaccination. Cohort A) symptomatic patients with clinical signs or symptoms suggestive of myocardial injury and Cohort B) asymptomatic patients without symptoms suggestive of myocardial injury who have had prior cardiac MRI.
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A - Symptomatic (Other): Those with clinical findings suggestive of myocarditis/myocardial injury after COVID-19 vaccination
  Interventions: Diagnostic Test: Cardiac PET/MRI; Diagnostic Test: Blood Biomarkers
- Cohort B - Asymptomatic (Other): Those without signs or symptoms suggestive of myocarditis after COVID-19 vaccination
  Interventions: Diagnostic Test: Cardiac PET/MRI; Diagnostic Test: Blood Biomarkers

INTERVENTIONS:
Diagnostic Test: Cardiac PET/MRI — An imaging technique that combines the strengths of both MRI and PET into one comprehensive study. This technique allows for detailed myocardial tissue characterization with MRI (including assessment of myocardial edema and fibrosis) and metabolic changes (including myocardial inflammation).
Diagnostic Test: Blood Biomarkers — Markers of cardiac damage, inflammation, circulating microRNA profiles, and COVID antibody levels will be evaluated in patients after COVID-19 vaccination.

SUMMARY:
The study will focus on cardiac blood and imaging biomarkers to facilitate early recognition of patients at risk for myocardial injury after COVID-19 vaccination. Ultimately, the intention is to identify patients at risk, reduce adverse events, and determine the need for longer-term follow-up in patients with myocardial injury after vaccination.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) vaccination frequently leads to minor side effects that may be more intense after the second dose, including fatigue and pain. However, there are emerging reports of more serious side effects in a minority of patients including myocarditis. Given the recent introduction of COVID-19 vaccination, there is limited understanding of: (i) prevalence and pattern of myocardial injury post vaccination, (ii) the risk factors for myocardial injury and adverse cardiac events post vaccination, and (iii) imaging and blood biomarkers for early recognition of patients at risk of adverse outcomes.

This study will address the above-mentioned knowledge gaps by focusing on patients who have received at least one dose of a COVID-19 vaccine. The study will focus on cardiac blood and imaging biomarkers to facilitate early recognition of patients at risk for myocardial injury after COVID-19 vaccination. Ultimately, the intention is to identify patients at risk, reduce adverse events, and determine the need for longer-term follow-up in patients with myocardial injury after vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 17 years (both Cohort A and B)
2. Received at least one dose of a COVID-19 vaccine in the past 6 months (both Cohort A and B)
3. Developed new clinical signs or symptoms suggestive of myocarditis/myocardial injury within one month of COVID vaccine administration without other known cause (Cohort A, only)

Exclusion Criteria:

1. Contraindications to cardiac PET/MRI
2. Current history of COVID-19

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of myocardial inflammation on PET/MRI | 6months and 12months
  The prevalence of myocardial inflammation on PET/MRI will be compared between symptomatic and asymptomatic patients

SECONDARY OUTCOMES:
Major adverse cardiac events (MACE) | 6months and 12months
  Defined as a composite of:
  1. Arrhythmias - new atrial or ventricular arrhythmia
  2. Acute coronary syndrome
     1. Acute myocardial infarction
     2. Unstable angina requiring revascularization (PCI or CABG)
  3. Heart failure hospitalization
  4. Cardiovascular death
Left ventricular dysfunction | 6months and 12months
  Defined as Left Ventricular Ejection Fraction (LVEF) < lower limit of normal on MRI
Myocardial edema | 6months and 12months
  Defined as high T2 > upper limit of normal on MRI

CONTACTS AND LOCATIONS:
Overall Officials: Kate Hanneman, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marschner CA, Thavendiranathan P, Gustafson D, Howe KL, Fish JE, Iwanochko RM, Wald RM, Abdel-Qadir H, Epelman S, Cheung AM, Hong R, Hanneman K. Myocardial Inflammation on FDG PET/MRI and Clinical Outcomes in Symptomatic and Asymptomatic Participants after COVID-19 Vaccination. Radiol Cardiothorac Imaging. 2023 Mar 9;5(2):e220247. doi: 10.1148/ryct.220247. eCollection 2023 Apr. PMID 36987440